CLINICAL TRIAL: NCT01642797
Title: Confocal Laser Endomicroscopy for the Diagnosis of Gastric Intestinal Metaplasia, Intraepithelial Neoplasia, and Carcinoma: A Multicenter, Randomized, Controlled Trial
Brief Title: Confocal Laser Endomicroscopy for the Diagnosis of Gastric Intestinal Metaplasia, Intraepithelial Neoplasia, and Carcinoma
Status: Unknown | Phase: Not Applicable | Type: Interventional
Last Known Status: Not yet recruiting
Sponsor: Shandong University (Other)
Collaborators: Prince of Wales Hospital, Shatin, Hong Kong (Other); National University Hospital, Singapore (Other); The University of New South Wales (Other)
Responsible Party: Principal Investigator, Yanqing Li, Chief of the department of Gastroenterology, Shandong University
Allocation: Randomized | Model: Parallel | Masking: Triple | Purpose: Diagnostic
Other Study IDs: 20120621
Record Dates: First submitted 2012-07-11; First posted 2012-07-17 (Estimated); Last update posted 2012-07-18 (Estimated); Status verified 2012-07

CONDITIONS: Gastric Intestinal Metaplasia; Gastric Intraepithelial Neoplasia; Gastric Carcinoma
Keywords: confocal laser endomicroscopy; gastric intestinal metaplasia; gastric intraepithelial neoplasia; gastric carcinoma
MeSH Terms: conditions — Stomach Neoplasms

STUDY DESIGN:
Who Masked: Participant, Investigator, Outcomes Assessor
Oversight: Data Monitoring Committee: Yes

ARMS (2):
- CLE-TB (Experimental): Confocal laser endomicroscopy with Targeted Biopsy
  Interventions: Device: Confocal laser endomicroscopy (Pentax, EG3870K)
- WLE-SB (Experimental): Standard White-light endoscopy with Standard Biopsy
  Interventions: Device: Standard White-light endoscopy (Pentax, 90i)

INTERVENTIONS:
Device: Confocal laser endomicroscopy (Pentax, EG3870K) — Confocal laser endomicroscopy with Targeted Biopsy
  Arms: CLE-TB
Device: Standard White-light endoscopy (Pentax, 90i) — Standard White-light endoscopy with Standard Biopsy
  Arms: WLE-SB

SUMMARY:
i. To determine whether Confocal Laser Endomicroscopy (CLE) with optical biopsy and targeted mucosal biopsy improves the diagnostic yield of gastric IM/IN/CA in high risk populations compared to WLE with standard biopsy protocol.

ii. To determine whether CLE with optical biopsy and targeted biopsy, as compared to WLE with standard biopsy, can reduce the number of biopsies needed per patient for detection of gastric IM/IN/carcinoma without the loss of corresponding diagnostic yield.

iii. To compare the sensitivity and specificity of CLE with WLE for the detection of gastric IM/IN/CA.

DETAILED DESCRIPTION:
Gastric cancer remains the world's second leading cause of cancer-related deaths. The prognosis for patients with this cancer clearly depends on stage at diagnosis. At least for the intestinal subtype of gastric adenocarcinoma, a cascade of histopathologic lesions has been defined: chronic gastritis, atrophic chronic gastritis, intestinal metaplasia (IM), and intraepithelial neoplasia (IN). The identification of these lesions and follow-up of patients in whom they are found could lead to diagnosis of gastric cancer at an early stage, thus improving patients' survival. The diagnosis of these lesions, which often appear in flat mucosa, is currently based on histopathologic examination of endoscopic biopsy specimens. However, conventional white-light endoscopy (WLE) for this purpose has high interobserver variability and a poor correlation with histopathologic finding.

Confocal laser endomicroscopy (CLE), producing both conventional WLE and confocal microscopic images, can provide a direct histological observation of the in vivo tissue without the need for biopsy. Recently, CLE has shown its value for diagnosing gastric IM, intraepithelial neoplasia and carcinoma. However, none of those CLE criteria for gastric IM, IN or carcinoma (CA) has been validated in various endoscopic centers, hence reducing the reliability and clinical application of them.

ELIGIBILITY:
Inclusion Criteria:

* Male or Female aged 18-80
* Patients with H. pylori infection, or histologically verified gastric intestinal metaplasia, low-grade intraepithelial neoplasia, and atrophic gastritis

Exclusion Criteria:

* Patients with gastrectomy, acute GI bleeding, and advanced gastric cancer
* Patients under conditions unsuitable for performing CLE including coagulopathy, impaired renal function, pregnancy or breastfeeding, and known allergy to fluorescein sodium
* Inability to provide informed consent and other situations that could interfere with the examination protocol

Ages: 18 Years to 80 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 242 (Estimated)
Dates: Start 2012-08; Primary Completion 2013-08 (Estimated); Study Completion 2013-09 (Estimated)

PRIMARY OUTCOMES:
number of participant with gastric IM/IN/CA | 1 year
  To determine whether CLE with optical biopsy and targeted mucosal biopsy improves the diagnostic yield of gastric IM/IN/CA in high risk populations compared to WLE with standard biopsy protocol.

SECONDARY OUTCOMES:
number of biopsies needed per patient | 1 year
  To determine whether CLE with optical biopsy and targeted biopsy, as compared to WLE with standard biopsy, can reduce the number of biopsies needed per patient for detection of gastric IM/IN/CA without the loss of corresponding diagnostic yield.

CONTACTS AND LOCATIONS:
Locations (4):
- the University of New South Wales, Bankstown-Lidcombe Hospital, Bankstown, Australia
- China (2):
  - the Prince of Wales Hospital, Chinese University of Hong Kong, Hong Kong, Hongkong
  - Qilu Hospital, Shandong University, Jinan, Shandong
- National University Hospital, National University of Singapore, Singapore, Singapore